CLINICAL TRIAL: NCT03019094
Title: Safety and Performance of the BlueWind RENOVA™ System for the Treatment of Patients Diagnosed With Overactive Bladder (OAB) (OPTIMIST-1 - Overactive Bladder Posterior Tibial Implantable MIcro STimulator - 1)
Brief Title: Overactive Bladder Posterior Tibial Implantable MIcro STimulator - 1
Acronym: OPTIMIST-1
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BlueWind Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G01-CLP-0001
Record Dates: First submitted 2017-01-05; First posted 2017-01-12 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; urge urinary incontinence; urgency frequency
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Implantation of the RENOVA tibial nerve stimulation system
  Interventions: Device: The RENOVA tibial nerve stimulation system

INTERVENTIONS:
Device: The RENOVA tibial nerve stimulation system — Study participants will be implanted with the RENOVA tibial nerve stimulation system

SUMMARY:
Interventional, Prospective, Open Label study

DETAILED DESCRIPTION:
Generally, subjects will be followed at 1, 2, 3, 4, 6, 9 and 12-months after activation with the RENOVA System.

The study will be conducted according the following phases:

* Recruitment, baseline assessment and compatibility test: Subjects fulfilling all inclusion and none of the exclusion criteria will be enrolled to the trial. Study candidates will sign an informed consent form, complete a standard 3-Day voiding diary, a quality of life questionnaire and global response assessment. Beck Depression Inventory II and General quality of life questionnaires will be completed in selected geographies. Study eligible subjects that have not experienced Posterior Tibial Nerve Stimulation treatment in the past will undergo a compatibility test to assure proper nerve conductivity. Data collected will serve as baseline.
* Implantation: Patients with positive response to the compatibility test (or that received Posterior Tibial Nerve Stimulation treatment in the past) will undergo unilateral implantation 4±1 weeks following recruitment with the BlueWind RENOVA System. Intra-operative sensory/motor response will be tested to confirm accurate location of the implant.
* Sensation assessment and activation: After a recovery period of approximately 30±7 days, subjects will complete a Brief 3-Day voiding diary and a quality of life questionnaire and a sensation assessment will be conducted: subjects will undergo an acute stimulation session of the tibial nerve to evaluate their sensory reaction to stimulation and parameters setting will be performed according to their individual sensations. Eventually, patients will be trained for system home use treatment. Therapy will be delivered daily for a minimum of 30 minutes once a day and maximum of 1 hour per day (in 2 sessions of 30 minutes), per physician discretion. Following activation of the device, patient will complete Brief 3-day voiding diaries once a week until the 1 month follow-up visit.
* Follow-ups (1-, 2-, and 3-months post-device activation): A 3-Day voiding diary and QoL questionnaire will be collected (brief 3-Day diaries on 1-, and 2-months follow up visits; and a 3-Day standard voiding diary on the 3-month follow up). Global Response Assessment and Beck Depression Inventory II will be collected on the 3-month follow-up visit (Beck Depression Inventory in selected geographies). Stimulation parameters will be checked and adjusted as needed by: (a) changing current amplitude; and/or (b) changing stimulation frequency; and/or changing pulse width; and/or (c) changing the number of daily treatment sessions. Location of paresthesia will be recorded in each of the clinic visits. The visit at 2 months will be performed by phone call to assess the patient status. Clinic visit may be followed at the discretion of the clinical team.
* Continued follow-ups: All subjects in the trial will undergo 4 additional visits (at 4-, 6- ,9- and 12-months post-device activation) until the end of the study at the 12-month visit. Similar to the visit at 2 months, the visit at 4 months will be performed by phone call to assess the patient status. Clinic visit may be followed at the discretion of the clinical team. Three-Day voiding diary, Quality of Life questionnaire, Global Response Assessment and Beck Depression Inventory II and General quality of life questionnaires (at selected geographies) will be collected at each of those visits (except for the 4- and 9-months visit in which only a 3-Day Brief voiding diary will be collected). General quality of life questionnaire will be completed at the 12-month visit in selected geographies. Stimulation parameters will be checked and adjusted as needed. Location of paresthesia will be recorded in each of the clinic visits

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Patient who is mentally competent with the ability to understand and comply with the requirements of the study.
3. Patient agrees to attend all follow-up evaluations and is willing to completely and accurately fill out voiding diaries and questionnaires, and is willing to complete required exams and tests.
4. Patients with overactive bladder symptoms including:

   * Urinary frequency greater than or equal to 8 voids/24 hours and less than 16 voids/24 hours AND/OR
   * Urinary urge incontinence of at least 2 incontinence episodes on a 3-Day voiding diary
5. If used, patients should be on stable dose of antimuscarinics and/or beta-3 adrenergic agonists for at least 6 weeks prior to enrollment and agree not to change their dose until the 3-month follow-up visit.
6. If used, patients should be on a stable dose of tricyclic antidepressants and Flomax for at least 6 weeks prior to enrollment and agree not to change their dose until the 3-month follow-up visit.
7. Patient who has failed conservative treatments after at least 6 months of treatment (i.e. lifestyle modification-fluid consumption, behavioral modification, and pharmacological therapy).
8. Patients with no clinical evidence of a tibial motor sensory deficit.
9. Patients with competent sphincter mechanism.
10. Patients with normally functioning upper urinary tract and no renal failure.
11. Leg circumference in the range of 20-30 cm at implantation site.
12. Patients with a standard 3-Day voiding diary at baseline.

Exclusion Criteria:

1. Previous participation in another study with any investigational drug or device within the past 90 days.
2. Any metal or other implant in the area of BlueWind RENOVA implantation site.
3. Patients who have not had stable OAB medications for at least 6 weeks.
4. Patients with neurogenic bladder.
5. Patients who are taking diuretics.
6. Patients who have received botulinum toxin injections within the past 12 months.
7. Patients who have received or are receiving nerve stimulation therapies for OAB treatment, including Sacral Nerve Stimulation (and are still implanted) or Posterior Tibial Nerve Stimulation (during the last 3 months).
8. Current pregnancy or attempting to get pregnant.
9. Previous urinary incontinence surgery or implantation of artificial graft material.
10. Any spinal or genitourinary surgery within the last 6 months.
11. Previous abdominoperineal resection of the rectum or radical hysterectomy (female)/ prostatectomy (male).
12. Skin, orthopedic or neurologic anatomical limitations that preclude implantation or/and use of the device.
13. Pelvic pain disorders.
14. Obvious clinically demonstrated genuine stress incontinence including mixed incontinence.
15. Any neurological disease or disorder including Alzheimer's, Parkinson, Multiple Sclerosis, neuropathy or injury resulting in neuropathy.
16. Current or recurrent urinary tract infection (3 or more infections in the last 6 months), or urinary tract obstruction such as benign prostatic hypertrophy, cancer, urethral stricture or presence of urinary stone.
17. History of Pelvic radiotherapy and chemotherapy.
18. Severe uncontrolled diabetes.
19. Patients anticipating magnetic resonance imaging (MRI) exams that are not allowed in the device labeling.
20. Presence of cystocele, enterocele or rectocele of grade 2 or more.
21. Patients with a documented history of allergic response to Platinum iridium, Titanium, Zirconia and Parylene.
22. Another active implant.
23. Have a life expectancy of less than 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse events | 6 and 12 months post-activation
  Incidence of serious adverse events (system and/or procedure related events)
Clinical improvement in urge urinary incontinence | 3 months post-activation
  Change from baseline in number of leaking episodes per day
Clinical improvement urinary frequency | 3 months post-activation
  Change from baseline in number of voids per day
Clinical improvement in degree of urgency | 3 months post-activation
  Change from baseline in degree of urgency prior to void

SECONDARY OUTCOMES:
Change in number of leaking episodes | 6- and 12 months post activation
  Change from baseline in number of leaking episodes
Change in number of voids | 6- and 12 months post activation
  Change from baseline in number of voids
Change in degree of urgency prior to void | 6- and 12 months post activation
  Change from baseline in degree of urgency prior to void
Change in number of absorbent pads | 3, 6, and 12 months post activation
  Change from baseline in number of Absorbent pads used due to leaking/day
Change in volume voided per void | 3, 6, and 12 months post activation
  Change from baseline of Volume voided/void
Change in urge urinary incontinence episodes | 3, 6, and 12 months post activation
  Change from baseline in severity of leaking episodes
Change in Quality of Life | 3, 6, and 12 months post activation
  Change from baseline in quality of life
Change in Global response of patient to treatment | 3, 6, and 12 months post activation
  Change from baseline in global response assessment
Change in Depression indices | 3, 6, and 12 months post activation
  Change from baseline in Beck Depression Inventory II